CLINICAL TRIAL: NCT06236997
Title: Adebrelimab and Concurrent Radiochemotherapy as First-line Treatment for Extensive-stage Small-cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-II-011
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-10

CONDITIONS: Small Cell Lung Carcinoma
Keywords: ES-SCLC; Concurrent Radiochemotherapy; Adebrelimab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Radiotherapy; EC regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (etoposide, carboplatin, radiation, Adebrelimab) (Experimental): Participants receive etoposide 100mg/m2 day1-3+carboplatin AUC 5 day 1(EC) combined with Adebrelimab（ PD-L1 inhibitor）1200mg day1 Q3w for 2 cycles, and the efficacy is evaluated 3 weeks after the treatment. If the efficacy evaluation is SD/PR/CR, concurrent radiotherapy(45Gy /3Gy/qd/3w) with EC(2 cycles) + Adebrelimab will be initiated. After concurrent chemoradiotherapy+ Adebrelimab, Adebrelimab was maintained until PD or intolerance or for at most 2 years.
  Interventions: Drug: Adebrelimab; Radiation: Radiation Therapy; Drug: etoposide, carboplatin(EC)

INTERVENTIONS:
Drug: Adebrelimab — Etoposide 100mg/m2 day1-3+carboplatin AUC 5 day 1(EC) combined with Adebrelimab（ PD-L1 inhibitor）1200mg day1 Q3w for 2 cycles, and the efficacy is evaluated 3 weeks after the treatment. If the efficacy evaluation is SD/PR/CR, concurrent radiotherapy(45Gy /3Gy/qd/3w) with EC(2 cycles) + Adebrelimab will be initiated. After concurrent chemoradiotherapy+ Adebrelimab, Adebrelimab was maintained until PD or intolerance or for at most 2 years.
Radiation: Radiation Therapy — Etoposide 100mg/m2 day1-3+carboplatin AUC 5 day 1(EC) combined with Adebrelimab（ PD-L1 inhibitor）1200mg day1 Q3w for 2 cycles, and the efficacy is evaluated 3 weeks after the treatment. If the efficacy evaluation is SD/PR/CR, concurrent radiotherapy(45Gy /3Gy/qd/3w) with EC(2 cycles) + Adebrelimab will be initiated. After concurrent chemoradiotherapy+ Adebrelimab, Adebrelimab was maintained until PD or intolerance or for at most 2 years.
Drug: etoposide, carboplatin(EC) — Etoposide 100mg/m2 day1-3+carboplatin AUC 5 day 1(EC) combined with Adebrelimab（ PD-L1 inhibitor）1200mg day1 Q3w for 2 cycles, and the efficacy is evaluated 3 weeks after the treatment. If the efficacy evaluation is SD/PR/CR, concurrent radiotherapy(45Gy /3Gy/qd/3w) with EC(2 cycles) + Adebrelimab will be initiated. After concurrent chemoradiotherapy+ Adebrelimab, Adebrelimab was maintained until PD or intolerance or for at most 2 years.

SUMMARY:
Patients with extensive-stage small-cell lung cancer (ES-SCLC) have poor prognosis, with limited treatment options. Chemo-immunotherapy is the standard 1st-line therapy for patients with ES-SCLC.When 4 cycles of etoposide+carboplatin (EC) or etoposide+cisplatin(EP) chemotherapy combined with PD-L1 inhibitor are effective, guidelines recommend additional thoracic radiotherapy.

In this study, the investigators bring radiotherapy forward, which means that after 2 cycles of EC chemotherapy plus Adebrelimab, participants with response（PR/CR/SD）will receive concurrent radiotherapy and 2 cycles of EC chemotherapy plus Adebrelimab, then maintenance therapy with Adebrelimab （Q3W）.

The purpose of this study is to explore the safety and efficacy of Adebrelimab combined with concurrent chemoradiotherapy in untreated participants with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
Participants receive EC chemotherapy combined with Adebrelimab for 2 cycles, and the efficacy will be evaluated. If the efficacy evaluation is SD/PR/CR, concurrent chemoradiotherapy combined with EC(2 cycles) + Adebrelimab will be initiated. After concurrent chemoradiotherapy + Adebrelimab, Adebrelimab was maintained until PD or intolerance or for at most 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Histologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system) ;
3. Must sign a written informed consent form prior to any study specific procedures;
4. No prior treatment for ES-SCLC;
5. No more than 5 lesions (including metastases),and at least one measurable lesion that meets RECIST 1.1 evaluation criteria;
6. Life expectancy more than 3 months;
7. ECOG PS 0-1

Exclusion Criteria:

1. Previous treatment with radiochemotherapy for limited-stage small cell lung cancer;
2. Subjects who previously received systemic antitumor or Immune checkpoint inhibitor therapy ;
3. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment;
4. Active brain metastases, Leptomeningeal metastasis(untreated central nervous system (CNS) metastases unless asymptomatic and lesion size<1cm;
5. Patients with spinal cord compression;
6. Patients with multiple liver metastases(except isolated lesion and lesion size<2cm);
7. Uncontrollable third cavity effusion (e.g. a large amount of pleural effusion, ascites, or pericardial effusion, etc.) requiring repeated drainage, which was judged by the investigator to be unsuitable for study;
8. The investigator judges that there are any patients who endanger the patient's safety, interfere with the study assessment, and have poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
6-m PFS rate | 6 months
  6-m PFS rate is defined as the percentage of participants whose disease is still progression-free at the 6th month

SECONDARY OUTCOMES:
ORR | up to 24 months.
  Objective response rate is defined as the proportion of subjects who have a CR or a PR
PFS | From date of the first treatment to the first documented disease progression, assessed up to 24 months
  Progression-free survival is defined as the time from the first treatment to the first documented disease progression
OS | From date of the first treatment to death due to any cause, assessed up to 24 months
  Overall survival is defined as the time from the first treatment to death due to any cause.
12-m PFS rate | 12 months
  12-m PFS rate is defined as the percentage of participants whose disease is still progression-free at the 12th month
AEs | up to 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qimig Wang, Doctor, Principal Investigator — Henan Cancer Hospital; Guangyuan Hu, Doctor, Principal Investigator — Tongji Hospital
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei